CLINICAL TRIAL: NCT00244569
Title: Development of a Breath Test for Monitoring Liver Metabolic Function in Patients With Chronic Liver Disease and Cirrhosis
Brief Title: Development of a Breath Test for Monitoring Patients With Liver Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Oridion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OBID-2005-VCU
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Fatty Liver; Cirrhosis
Keywords: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; Liver Function; Metabolism; Cirrhosis; Fibrosis; Liver
MeSH Terms: conditions — Fatty Liver; Fibrosis; Non-alcoholic Fatty Liver Disease

INTERVENTIONS:
Drug: 13C-Methacetin
Device: Breath ID Machine

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the Oridion Breath ID machine in monitoring liver metabolic functions.

DETAILED DESCRIPTION:
Percutaneous liver biopsy has been utilized for decades to assess the severity of chronic liver disease, regardless of etiology. During this procedure a core sample of liver is obtained and examined histologically for the presence of inflammation, fibrosis and other features characteristic of specific liver disorders.Although liver biopsy is the gold standard by which to assess liver disease severity the procedure has significant limitations. Liver biopsy is a costly, invasive procedure with risks for morbidity and mortality. In addition, liver biopsy and examination of liver histology is subject to sampling variation and the manner by which these findings are evaluated and reported by individual pathologists.

Because of these limitations several investigators have attempted to develop alternative methods by which to assess liver disease severity. One approach was the development of serum markers which can estimate liver fibrosis. Such tests were developed by analyzing a battery of serum liver chemistries and the platelet count. Unfortunately, the test cannot detect more subtle changes in liver fibrosis and does not provide any information regarding hepatic function in patients with established cirrhosis. The concept of a metabolic liver function test, which could be utilized to assess the liver function was first explored several decades ago (20). Such tests are performed by administering a compound either orally or intravenously. The compound is removed by the liver from the blood, metabolized and a metabolic product is released back into the blood and excreted in the urine, saliva or exhaled breath; or the metabolic product is excreted in bile. Measuring the amount of the administered product that remains in serum over time or the amount of metabolic product which is produced and/or the rate at which this product is excreted provides an accurate measure of hepatic metabolic function.

Breath testing utilizing 13C labeled substrates provides a safe, non-invasive means for measuring hepatic metabolism. 13C is a stable, non-radioactive isotope which can be incorporated into a specific location within a test substrate so that it would be released when the compound is metabolized by the liver. Ideally, the 13C-compound would be administered orally, rapidly absorbed, metabolized by the liver and 13CO2 would be measured in exhaled breath within 20-30 minutes. Hepatic metabolism of the compound would be assessed by measuring the ratio of 13C/12C in exhaled breath. The ability to detect, differentiate and quantify 13C and 12C in exhaled CO2 has been greatly facilitated by the recent development of the Breath ID® collection system and analyzer unit. This portable device continuously senses exhaled breath and analyzes CO2 in real-time through a nasal cannula worn by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (age 18+)
* Liver histology consistent with NAFLD/NASH performed within the past 24 months
* Patients with cirrhosis must have ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI) examination of liver performed within the previous 6 months demonstrating no evidence for hepatocellular carcinoma

Exclusion Criteria:

* Any liver disease beyond NAFLD/NASH
* Severe congestive heart failure
* Severe pulmonary hypertension
* Chronic renal insufficiency defined by a serum creatinine above normal
* Uncontrolled diabetes mellitus
* Any autoimmune disorder which is currently being treated with immune suppressive medication
* Proven or suspected hepatocellular carcinoma
* Previous surgical bypass surgery for morbid obesity
* Extensive small bowel resection
* Patients currently receiving total parenteral nutrition
* Recipients of any organ transplant
* Women who are pregnant
* Patients who, in the opinion of the investigator, should not be enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The mean and standards of results obtained from the Breath ID system for each of the 3 groups of patients with nonalcoholic fatty liver disease/nonalcoholic steatohepatitis (NAFLD/NASH) will be compared by chi squared analysis.
A p value of 0.05 or less will be considered significant.

SECONDARY OUTCOMES:
Receiver-operator curves will be developed to compare the results of the Breath ID to each histologic group of patients studied. A p value of 0.05 will be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell L. Shiffman, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Ludwig J, Dickson ER, McDonald GS. Staging of chronic nonsuppurative destructive cholangitis (syndrome of primary biliary cirrhosis). Virchows Arch A Pathol Anat Histol. 1978 Aug 22;379(2):103-12. doi: 10.1007/BF00432479. No abstract available. PMID 150690
- [Background] Ludwig J, Barham SS, LaRusso NF, Elveback LR, Wiesner RH, McCall JT. Morphologic features of chronic hepatitis associated with primary sclerosing cholangitis and chronic ulcerative colitis. Hepatology. 1981 Nov-Dec;1(6):632-40. doi: 10.1002/hep.1840010612. PMID 7308996
- [Background] Richard S, Guerret S, Gerard F, Tebib JG, Vignon E. Hepatic fibrosis in rheumatoid arthritis patients treated with methotrexate: application of a new semi-quantitative scoring system. Rheumatology (Oxford). 2000 Jan;39(1):50-4. doi: 10.1093/rheumatology/39.1.50. PMID 10662873
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461
- [Background] Knodell RG, Ishak KG, Black WC, Chen TS, Craig R, Kaplowitz N, Kiernan TW, Wollman J. Formulation and application of a numerical scoring system for assessing histological activity in asymptomatic chronic active hepatitis. Hepatology. 1981 Sep-Oct;1(5):431-5. doi: 10.1002/hep.1840010511. PMID 7308988
- [Background] Ishak KG. Pathologic features of chronic hepatitis. A review and update. Am J Clin Pathol. 2000 Jan;113(1):40-55. doi: 10.1309/42D6-W7PL-FX0A-LBXF. PMID 10631857
- [Background] Scheuer PJ, Ashrafzadeh P, Sherlock S, Brown D, Dusheiko GM. The pathology of hepatitis C. Hepatology. 1992 Apr;15(4):567-71. doi: 10.1002/hep.1840150402. PMID 1551631
- [Background] Bedossa P, Poynard T. An algorithm for the grading of activity in chronic hepatitis C. The METAVIR Cooperative Study Group. Hepatology. 1996 Aug;24(2):289-93. doi: 10.1002/hep.510240201. PMID 8690394
- [Background] McGill DB, Rakela J, Zinsmeister AR, Ott BJ. A 21-year experience with major hemorrhage after percutaneous liver biopsy. Gastroenterology. 1990 Nov;99(5):1396-400. doi: 10.1016/0016-5085(90)91167-5. PMID 2101588
- [Background] Perrault J, McGill DB, Ott BJ, Taylor WF. Liver biopsy: complications in 1000 inpatients and outpatients. Gastroenterology. 1978 Jan;74(1):103-6. PMID 618417
- [Background] Janes CH, Lindor KD. Outcome of patients hospitalized for complications after outpatient liver biopsy. Ann Intern Med. 1993 Jan 15;118(2):96-8. doi: 10.7326/0003-4819-118-2-199301150-00003. PMID 8416324
- [Background] Ratziu V, Charlotte F, Heurtier A, Gombert S, Giral P, Bruckert E, Grimaldi A, Capron F, Poynard T; LIDO Study Group. Sampling variability of liver biopsy in nonalcoholic fatty liver disease. Gastroenterology. 2005 Jun;128(7):1898-906. doi: 10.1053/j.gastro.2005.03.084. PMID 15940625
- [Background] Fontana RJ, Lok AS. Noninvasive monitoring of patients with chronic hepatitis C. Hepatology. 2002 Nov;36(5 Suppl 1):S57-64. doi: 10.1053/jhep.2002.36800. PMID 12407577
- [Background] Soloway RD, Baggenstoss AH, Schoenfield LJ, Summerskill WH. Observer error and sampling variability tested in evaluation of hepatitis and cirrhosis by liver biopsy. Am J Dig Dis. 1971 Dec;16(12):1082-6. doi: 10.1007/BF02235164. No abstract available. PMID 5135770
- [Background] Regev A, Berho M, Jeffers LJ, Milikowski C, Molina EG, Pyrsopoulos NT, Feng ZZ, Reddy KR, Schiff ER. Sampling error and intraobserver variation in liver biopsy in patients with chronic HCV infection. Am J Gastroenterol. 2002 Oct;97(10):2614-8. doi: 10.1111/j.1572-0241.2002.06038.x. PMID 12385448
- [Background] Poynard T, McHutchison J, Manns M, Myers RP, Albrecht J. Biochemical surrogate markers of liver fibrosis and activity in a randomized trial of peginterferon alfa-2b and ribavirin. Hepatology. 2003 Aug;38(2):481-92. doi: 10.1053/jhep.2003.50319. PMID 12883493
- [Background] Rosenberg WM, Voelker M, Thiel R, Becka M, Burt A, Schuppan D, Hubscher S, Roskams T, Pinzani M, Arthur MJ; European Liver Fibrosis Group. Serum markers detect the presence of liver fibrosis: a cohort study. Gastroenterology. 2004 Dec;127(6):1704-13. doi: 10.1053/j.gastro.2004.08.052. PMID 15578508
- [Background] Poynard T, Imbert-Bismut F, Munteanu M, Messous D, Myers RP, Thabut D, Ratziu V, Mercadier A, Benhamou Y, Hainque B. Overview of the diagnostic value of biochemical markers of liver fibrosis (FibroTest, HCV FibroSure) and necrosis (ActiTest) in patients with chronic hepatitis C. Comp Hepatol. 2004 Sep 23;3(1):8. doi: 10.1186/1476-5926-3-8. PMID 15387887
- [Background] Burra P, Masier A. Dynamic tests to study liver function. Eur Rev Med Pharmacol Sci. 2004 Jan-Feb;8(1):19-21. PMID 15209151
- [Background] Gadano A, Hadengue A, Vachiery F, Moreau R, Sogni P, Soupison T, Yang S, Cailmail S, Lebrec D. Relationship between hepatic blood flow, liver tests, haemodynamic values and clinical characteristics in patients with chronic liver disease. J Gastroenterol Hepatol. 1997 Feb;12(2):167-71. doi: 10.1111/j.1440-1746.1997.tb00401.x. PMID 9083919
- [Background] Bergstrom M, Soderman C, Eriksson LS. A simplified method to determine galactose elimination capacity in patients with liver disease. Scand J Clin Lab Invest. 1993 Nov;53(7):667-70. doi: 10.3109/00365519309092569. PMID 8272755
- [Background] Merkel C, Gatta A, Zoli M, Bolognesi M, Angeli P, Iervese T, Marchesini G, Ruol A. Prognostic value of galactose elimination capacity, aminopyrine breath test, and ICG clearance in patients with cirrhosis. Comparison with the Pugh score. Dig Dis Sci. 1991 Sep;36(9):1197-203. doi: 10.1007/BF01307508. PMID 1893804
- [Background] Jodynis-Liebert J, Flieger J, Matuszewska A, Juszczyk J. Serum metabolite/caffeine ratios as a test for liver function. J Clin Pharmacol. 2004 Apr;44(4):338-47. doi: 10.1177/0091270004263468. PMID 15051740
- [Background] Munoz AE, Miguez C, Rubio M, Bartellini M, Levi D, Podesta A, Niselman V, Terg R. Lidocaine and monoethylglycinexylidide serum determinations to analyze liver function of cirrhotic patients after oral administration. Dig Dis Sci. 1999 Apr;44(4):789-95. doi: 10.1023/a:1026630313038. PMID 10219840
- [Background] Lara Baruque S, Razquin M, Jimenez I, Vazquez A, Gisbert JP, Pajares JM. 13C-phenylalanine and 13C-methacetin breath test to evaluate functional capacity of hepatocyte in chronic liver disease. Dig Liver Dis. 2000 Apr;32(3):226-32. doi: 10.1016/s1590-8658(00)80825-7. PMID 10975773
- [Background] Festi D, Capodicasa S, Sandri L, Colaiocco-Ferrante L, Staniscia T, Vitacolonna E, Vestito A, Simoni P, Mazzella G, Portincasa P, Roda E, Colecchia A. Measurement of hepatic functional mass by means of 13C-methacetin and 13C-phenylalanine breath tests in chronic liver disease: comparison with Child-Pugh score and serum bile acid levels. World J Gastroenterol. 2005 Jan 7;11(1):142-8. doi: 10.3748/wjg.v11.i1.142. PMID 15609414
- [Background] Matsumoto K, Suehiro M, Iio M, Kawabe T, Shiratori Y, Okano K, Sugimoto T. [13C]methacetin breath test for evaluation of liver damage. Dig Dis Sci. 1987 Apr;32(4):344-8. doi: 10.1007/BF01296285. PMID 3030679
- [Background] Shiffman ML, Luketic VA, Sanyal AJ, Duckworth PF, Purdum PP 3rd, Contos MJ, Mills AS, Edinboro LE, Poklis A. Hepatic lidocaine metabolism and liver histology in patients with chronic hepatitis and cirrhosis. Hepatology. 1994 Apr;19(4):933-40. PMID 8138268
- [Background] Shiffman ML, Fisher RA, Sanyal AJ, Edinboro LE, Luketic VA, Purdum PP 3rd, Raymond P, Posner MP. Hepatic lidocaine metabolism and complications of cirrhosis. Implications for assessing patient priority for hepatic transplantation. Transplantation. 1993 Apr;55(4):830-5. doi: 10.1097/00007890-199304000-00028. PMID 8475560
- [Background] Adamek RJ, Goetze O, Boedeker C, Pfaffenbach B, Luypaerts A, Geypens B. 13C-methacetin breath test: isotope-selective nondispersive infrared spectrometry in comparison to isotope ratio mass spectrometry in volunteers and patients with liver cirrhosis. Z Gastroenterol. 1999 Dec;37(12):1139-43. PMID 10666836
- [Background] Klatt S, Taut C, Mayer D, Adler G, Beckh K. Evaluation of the 13C-methacetin breath test for quantitative liver function testing. Z Gastroenterol. 1997 Aug;35(8):609-14. PMID 9297776
- [Background] Myers J, Ahnve S, Froelicher V, Livingston M, Jensen D, Abramson I, Sullivan M, Mortara D. A randomized trail of the effects of 1 year of exercise training on computer-measured ST segment displacement in patients with coronary artery disease. J Am Coll Cardiol. 1984 Dec;4(6):1094-102. doi: 10.1016/s0735-1097(84)80127-8. PMID 6389645
- [Background] Petrolati A, Festi D, De Berardinis G, Colaiocco-Ferrante L, Di Paolo D, Tisone G, Angelico M. 13C-methacetin breath test for monitoring hepatic function in cirrhotic patients before and after liver transplantation. Aliment Pharmacol Ther. 2003 Oct 15;18(8):785-90. doi: 10.1046/j.1365-2036.2003.01752.x. PMID 14535871
- [Background] Ciccocioppo R, Candelli M, Di Francesco D, Ciocca F, Taglieri G, Armuzzi A, Gasbarrini G, Gasbarrini A. Study of liver function in healthy elderly subjects using the 13C-methacetin breath test. Aliment Pharmacol Ther. 2003 Jan;17(2):271-7. doi: 10.1046/j.1365-2036.2003.01413.x. PMID 12534413
- [Background] Krumbiegel P, Gunther K, Faust H, Mobius G, Hirschberg K, Schneider G. Nuclear medicine liver function tests for pregnant women and children. 1. Breath tests with 14C-methacetin and 13C-methacetin. Eur J Nucl Med. 1985;10(3-4):129-33. doi: 10.1007/BF00252720. PMID 3996441
- [Background] Krumbiegel P, Stolz L, Herbarth O, Braun W, Boehm G, Kausch S, Wirsing A. Is the [15N]methacetin liver function test suited to estimate environmental effects on the maturity of neonates? Cent Eur J Public Health. 1994 Jun;2(1):49-51. PMID 7812247